CLINICAL TRIAL: NCT02500264
Title: The Effect of Non Invasive Electrical Stimulation Therapy on Gastroesophageal Reflux Disease (GERD) Symptoms - Proof of Concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ram Dickman, Gastroenterologist, manager of the GI movement service in RMC, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0293-15-RMC
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Transcutaneous Electric Nerve Stimulation

ARMS (4):
- Protocol #1 (Active Comparator): interventions: 1.6Hz, Rampdown 0.4S, electrodes position - both L.Rectus Abdominis, 5cmX5cm Size, on inspirium
  Interventions: Device: TENS
- Protocol #2 (Active Comparator): 1Hz, Rampdown 0.6S, electrodes position - both Rectus Abdominis, 5cmX5cm Size, on inspirium
  Interventions: Device: TENS
- Protocol #3 (Active Comparator): 1.6Hz, Rampdown 0.4S, electrodes position - L.Rectus Abdominis and L.External Oblique, 5cmX5cm Size, on inspirium Oblique
  Interventions: Device: TENS
- Protocol #4 (Active Comparator): 1Hz, Rampdown 0.6S, electrodes position - L.Rectus Abdominis and L.External Oblique, 5cmX5cm Size, on inspirium
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS

SUMMARY:
The aims of the study: To evaluate whether the use of a specific TENS technology can improve GERD symptoms and esophageal acid exposure.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 episodes of heartburn and/or regurgitation in a week for at least 3 months.
* evidence for an abnormal esophagal acid exposure on impedance-pH monitoring (tested in the last 2 years off PPI)

Exclusion Criteria:

* gastric or esophagal surgery
* active peptic ulcer disease
* malignancy
* pregnancy
* uncontrolled diabetes mellitus
* severe cardiac conditions such as cardiac arrhythmia or ischemia or cardiac pacemaker/defibrillator
* allergy to adhesives/patches
* severe pulmonary disease
* obesity (BMI>30)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity questionnaire (heartburn and regurgitation) before and after treatment | 34 days

SECONDARY OUTCOMES:
Esophageal acid exposure before and after treatment | 34 days
  Ph monitoring

CONTACTS AND LOCATIONS:
Overall Officials: ram dickman, professor, Principal Investigator — MD
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel